CLINICAL TRIAL: NCT04746430
Title: COVID-19 Primary Care Platform for Early Treatment and Recovery (COPPER) Study: an Open-label Randomized Controlled Trial
Brief Title: COVID-19 Primary Care Platform for Early Treatment and Recovery (COPPER) Study
Acronym: COPPER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Too few patients
Sponsor: General Practitioners Research Institute (Network)
Collaborators: Huisartsenzorg Drenthe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPRI-21001-COV; 2021-000235-30 (EudraCT Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 6 mg dexamethasone prescribed during ten days and as a precaution combined with electronic monitoring of saturation and other signs and symptoms
  Interventions: Drug: Dexamethasone
- Control (No Intervention): Only remote monitoring

INTERVENTIONS:
Drug: Dexamethasone — 6 mg dexamethasone prescribed during ten days and as a precaution combined with electronic monitoring of saturation and other signs and symptoms
  Arms: Intervention

SUMMARY:
The COVID-19 coronavirus has led to a global pandemic of respiratory diseases with an increase in hospitalization and death risk. To keep COVID-19 manageable for healthcare, early treatment is urgently needed to avoid hospitalization. Dexamethasone can dampen the exaggerated cytokine response to COVID-19 and is a promising agent for preventing disease aggravation, hospitalization and death. However, the evidence on the effectiveness, safety and cost-effectiveness of dexamethasone treatment in primary care is inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* A positive test for SARS-CoV-2
* A GP consultation for deteriorating COVID-19 symptoms

Additional inclusion criteria in order to be eligible for randomization to the trial:

- Exercise-induced desaturation, defined as SpO2<92% (<90% for COPD patients) and/or an absolute drop of ≥4% in SpO2 after a 1-minute sit-to-stand test

OR

- SpO2<92% (<90% for COPD patients) in rest with GP's and patient's shared decision to keep patient at home despite this in itself being an indication for referral to hospital

Exclusion Criteria:

* Inability to understand and sign the written consent form
* Inability to perform saturation measurements or sit-to-stand test
* Not willing to be admitted to hospital
* On the discretion of the recruiting clinician if he or she deems a patient not eligible

The following criterion will be used to exclude patients from randomization to the trial:

* Contra-indication for dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Hospitalization/death | 28 days
  Time to first hospital admission or death

SECONDARY OUTCOMES:
Recovery | 28 days
  To assess the effectiveness of early treatment with dexamethasone in reducing time to recovery inpatients who are carefully monitored by their GP after a consultation for deteriorating COVID-19
Disease severity | 28 days
  To assess the effectiveness of early treatment with dexamethasone in reducing COVID-19 disease severity in patients who are remotely monitored by their GP after a consultation for deteriorating symptoms
HCRU | 28 days
  To assess the effectiveness of the intervention in reducing healthcare resource utilization (HCRU)

CONTACTS AND LOCATIONS:
Overall Officials: Janwillem Kocks, Prof, Principal Investigator — General Practitioners Research Institute
Locations (1):
- GPRI, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided